CLINICAL TRIAL: NCT04007432
Title: Nocturnal Hypoxia in Patients Hospitalized in Orthogeriatrics After Hip Fracture
Brief Title: Nocturnal Hypoxia in Geriatric Patients After Hip Fracture
Acronym: HIPOX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP190391; 2019-A01084-53 (Other: ANSM)
Record Dates: First submitted 2019-06-18; First posted 2019-07-05 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Delirium; Hypoxia
Keywords: nocturnal hypoxia; delirum developpement
MeSH Terms: conditions — Delirium; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Older patients with hip fracture (Experimental): Older patients admitted for hip fracture surgery
  Interventions: Other: pulse oxymeter

INTERVENTIONS:
Other: pulse oxymeter — Nocturnal oxymetry data will be continuously collected during nighttime by a pulse oxymeter, covering for 1 to 3 nights.

SUMMARY:
Delirium is a common complication following hip fracture surgery (HFS) in older people. Postoperative hypoxia has also been associated with delirium, but not specifically in geriatric patients. The aim of the study is to demonstrate that post-operative hypoxia is associated with in-hospital complications in patients with HFS.

DETAILED DESCRIPTION:
Patients hospitalized in orthogeriatric unit after HFS will be monitored for nocturnal SpO2 with a pulse oximeter continuously during 3 nights. In-hospital complications will be recorded prospectively in all patients, especially the occurrence of delirium with the CAM scale. The hypoxia vs non-hypoxia (more than 20% of the time spent with SpO2<90%) groups will be analyzed for clinical characteristics, comorbidities and medication use.

The statistical association between severe post-operative nocturnal hypoxemia and occurrence of delirium will be assessed. The dependance between this association and daytime SpO2 will also be assessed. The potential confirmation of an association between post-operative nocturnal hypoxemia in patients with HFS and the occurrence of delirium will lead the reflection on a clinical trial testing the benefit of oxygen therapy in the prevention of post-operative delirium, to improve the medical care of orthogeriatric patients.

ELIGIBILITY:
Inclusion Criteria:

* age over 70 years old,
* hospitalized in orthogeriatrics for hip fracture surgery
* information about the study and expression of non opposition
* Expected hospital stay of 5 nights or more

Exclusion Criteria:

* patient under guardianship,
* any other type of fracture associated,
* oxymetry recording not possible (behavioral disorders, night stirring,...)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2027-02-05 (Estimated); Study Completion 2027-02-05 (Estimated)

PRIMARY OUTCOMES:
Delirium | Month 1
  Delirum or not, diagnosed with CAM (Confusion Assessment Method). Association between nocturnal hypoxia and delirium will be study.

SECONDARY OUTCOMES:
In-hospital complications | Month 1
  Occurrence of in-hospital complications (infection, cardiac, etc). Association between nocturnal hypoxia and others medical complications (infection, cardiac, etc) will be study.
Length of hospitalisation stay in othogeriatrics unit | Month 1
  Length of stay in othogeriatrics unit. Association between nocturnal hypoxia and length of hospitalisation stay in othogeriatrics unit will be study.
walking status (functional status) | Month 1
  walking status (possible with/without help, wheelchair or bedridden) Association between nocturnal hypoxia and functional status will be study.
walking status (functional status) | Month 1
  walking status (possible with/without help, wheelchair or bedridden). Association between nocturnal hypoxia and functional status will be study.
walking speed (functional status) | Month 1
  walking speed for 5 meter. Association between nocturnal hypoxia and functional status will be study.
Physical performance (functional status) | Month 1
  Short Physical Performance Battery (SPPB) is an objective assessment tool for evaluating lower extremity functioning in older persons.
Dependency | Month 1
  Activities of Daily Living (ADL) and Instrumental Activities of Daily Living (IADL) are instrument to assess independent living skills.
  Association between nocturnal hypoxia and independent living skills will be study.
Dependency | Month 6
  Activities of Daily Living (ADL) and Instrumental Activities of Daily Living (IADL) are instrument to assess independent living skills.
  Association between nocturnal hypoxia and independent living skills will be study.
Mortality | Month 1
  Vital status will be raised
Mortality | Month 6
  Vital status will be raised
Nocturnal hypercapnia | Month 1
  Nocturnal hypercapnia defined by more than 10% time spent with a transcutaneous TcPCO2 ≥50mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Kiyoka KINUGAWA, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Service de gériatrie, Hopital Saint Antoine, Paris
  - Service de Gériatrie Hopital de La Pitié Salpetriere, Paris

IPD SHARING:
Plan to Share IPD: No